CLINICAL TRIAL: NCT01424072
Title: Applicability of Auriculotherapy as a Strategy for Stress and Coping in Nursing Professionals
Brief Title: Auriculotherapy as a Coping Strategy in Professional Nursing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonice Fumiko Sato Kurebayashi, Leonice Fumiko Sato Kurebayashi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 0060.0.198.000-09
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Stress, Psychological; Coping Behavior
Keywords: stress psychological; coping behavior
MeSH Terms: conditions — Stress, Psychological | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): Control Group didn't receive any treatment and was evaluated at the same time and the same way of interventions group
- Auriculotherapy by needles (Experimental): The investigators used 3 points, Shenmen, Kidney, and Brain Stem with semi-permanent needles of 1.8 mm, 1 time per week for 8 sessions.
  Interventions: Other: auriculotherapy by needles
- Auriculotherapy by seeds (Experimental): The investigators used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.
  Interventions: Other: auriculotherapy by seeds

INTERVENTIONS:
Other: auriculotherapy by needles — The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
  Other Names: auricular acupuncture
  Arms: Auriculotherapy by needles
Other: auriculotherapy by seeds — We used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.The subjects were instructed to stimulate the points three times a day.
  Other Names: auricular acupuncture by seeds
  Arms: Auriculotherapy by seeds

SUMMARY:
This randomized clinical trial aimed at evaluating the auriculotherapy as coping strategies in 75 nursing professionals in a University Hospital.

DETAILED DESCRIPTION:
There is consensus that psychological and social factors can lead to physical health problems of individuals and coping strategies in stressful situations may be crucial for the mental, physical and social development of people. Taking care of professionals who provide health services is a key strategy, since good results depend on the service, especially in work teams healthy and, therefore, able to promote the humanization of service.

ELIGIBILITY:
Inclusion Criteria:

* Average and high score by the List of Stress Symptoms
* Voluntary participation in the study
* Availability of time for submission to the sessions

Exclusion Criteria:

* Pregnancy
* Medical license or vacation during the period
* Low score of stress

Ages: 23 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonice FS Kurebayashi, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital Universitário de São Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted between January and September 2011 at University Hospital. Study participants were professionals from different sectors of the hospital after the invitation and 109 people answered the Stress Symptoms List. Obeying the exclusion criteria, 75 subjects were enrolled and randomized into three groups.
Pre-assignment Details: Of the 109 subjects, 4 were eliminated for having a low level of stress and three for not belonging to nursing staff.
Groups:
- Auriculotherapy by Needles: The investigators used 3 points, Shenmen, Kidney, and Brain Stem with semi-permanent needles of 1.8 mm, 1 time per week for 8 sessions.
  auriculotherapy by needles : The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
- Auriculotherapy by Seeds: The investigators used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.
  auriculotherapy by seeds : We used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.The subjects were instructed to stimulate the points three times a day.
Period: Overall Study
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Started | 27 | 26 | 22
Completed | 27 | 26 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group | Total
Number analyzed (Participants) | 27 | 26 | 22 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 22 | 75
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.37 (8.23) | 45.57 (6.40) | 39.25 (13.17) | 42.06 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 21 | 71
  Male | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Brazil | 27 | 26 | 22 | 75

OUTCOME MEASURES:

1. Secondary Outcome: Stress Scale
Description: Scale information: Stress Symptoms List (LSS)with 60 items (better outcome)Low score: 12/29 points; Medium score: 30/60 points; High score: 61/120 points; Very high score (worse outcome): >120 points.
Time Frame: after 60 days
Population: Of the 109 subjects, four were eliminated for having a low level of stress and three for not belonging to nursing staff;seven didn't appear in the first session. Some lost sessions and were also excluded. One abandoned the treatment because of the side effects, one didn't complete the questionnaire, seven went on vacation or sick leave(2).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Number analyzed (Participants) | 27 | 26 | 22
units on a scale | 59.84 (23.04) | 67.10 (23.77) | 67.87 (25.73)
Statistical Analysis 1: Comparison: Auriculotherapy by Needles vs Auriculotherapy by Seeds vs Control Group; The main objective was to compare the difference among the control group, seeds and needles and to recognize significant outcomes of auriculotherapy by seeds or needles; Test type: Superiority or Other; p = 0.023, ANOVA — It was verified the normality of data distribution and the homogeneity of variance

2. Primary Outcome: Coping Strategy: Domain Social Support(After 60 Days)
Description: Scale information: Folkman and Lazarus Coping Strategy Inventory with 66 items. The scale is constructed by 8 different "domains": confrontation, distancing, self-control, social support, acceptance of responsibility, escape avoidance, problem solving and positive reappraisal.The questions are scored by Likert scale: 0 (not used this strategy); 1 (used somewhat); 2 (used enough) and 3(used in large quantities) to the 66 items (Folkman and Lazarus Coping Strategy Inventory). It performed a summation of items and defined the scores: 0-4 points (not use this strategy), 5-9 (use this strategy a bit), 10-14 ( use this strategy quite) 14-18 (use strategy plenty).
Time Frame: after 60days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Number analyzed (Participants) | 27 | 26 | 22
units on a scale | 8.81 (2.50) | 8.73 (3.2) | 11.32 (4.3)
Statistical Analysis 1: Comparison: Auriculotherapy by Needles vs Auriculotherapy by Seeds vs Control Group; It was carried out the analysis of variance (ANOVA) among the groups in the 3rd assessment (after 60 days) and at the follow up (after 75 days). The main objective was to compare the difference among the control group, seeds and needles and to recognize significant outcomes of auriculotherapy by seeds or needles; Test type: Superiority or Other; p = 0,022, ANOVA — It was verified the normality of data distribution and the homogeneity of variance; This result was only to the domain Social Support

3. Primary Outcome: Coping Strategy: Distancing Domain
Description: The questions are scored by Likert scale: 0 (not used this strategy); 1 (used somewhat); 2 (used enough) and 3(used in large quantities) to the 66 items (Folkman and Lazarus Coping Strategy Inventory). It performed a summation of items and defined the scores: 0-4 points (not use this strategy), 5-9 (use this strategy a bit), 10-14 ( use this strategy quite) 14-18 (use strategy plenty).
Time Frame: after 75 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Number analyzed (Participants) | 27 | 26 | 22
units on a scale | 6.33 (1.34) | 6.65 (1.46) | 7.36 (2.32)
Statistical Analysis 1: Comparison: Auriculotherapy by Needles vs Auriculotherapy by Seeds vs Control Group; It was carried out the analysis of variance (ANOVA) among the groups at the follow up (after 75 days). The main objective was to compare the difference among the control group, seeds and needles and to recognize significant outcomes of auriculotherapy by seeds or needles; Test type: Superiority or Other; p = 0.039, ANOVA — It was verified the normality of data distribution and the homogeneity of variance
Statistical Analysis 2: Comparison: Auriculotherapy by Needles vs Auriculotherapy by Seeds vs Control Group; Coping Strategy: Confrontation domain; Test type: Superiority or Other; p = 0.029, ANOVA; It was carried out the analysis of variance (ANOVA) among the groups at the follow up and then it was used the post hoc test

4. Primary Outcome: Coping Strategy: Social Support Domain
Description: as for outcome 2
Time Frame: after 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Number analyzed (Participants) | 27 | 26 | 22
units on a scale | 8.81 (2.50) | 8.73 (3.2) | 11.32 (4.3)

ADVERSE EVENTS:
Time Frame: after 4 sessions (one month)
Description: The main symptoms or adverse events were:
  Nightmares; Complaints of anxiety and unrest; Anxiety for food; Itching and redness in the auricular points.
Arm/Group | Auriculotherapy by Needles | Auriculotherapy by Seeds | Control Group
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 3/27 | 1/26 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auriculotherapy by Needles (N=27) | Auriculotherapy by Seeds (N=26) | Control Group (N=22)
Nightmares (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Complaints of anxiety and unrest (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety for food (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Itching and redness in the auricular point (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Number of the participants(reduced sample)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The copyright of the search results are the exclusive property of Latin American Journal of Nursing, barring any reproduction, in whole or in part in any form or means of printed or electronic, without the prior and necessary authorization is requested.